CLINICAL TRIAL: NCT06892132
Title: A Randomized Control Trial of a Supervised Peanut Feeding Clinic to Increase Early Peanut Introduction
Brief Title: Evaluation of a Supervised Clinical Feeding Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Corinna Rea, Assistant Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P00050109
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Peanut Allergies in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Families will receive guidance about early peanut introduction via a handout.
  Interventions: Other: Handout
- Intervention (Experimental): Families will receive guidance about early peanut introduction via handout as well as a supervised feeding visit.
  Interventions: Other: Supervised feeding intervention

INTERVENTIONS:
Other: Supervised feeding intervention — Participants will be fed a peanut product during a supervised feeding visit and observed for an allergic reaction.
  Arms: Intervention
Other: Handout — Participants will receive a handout on how to introduce peanut products.
  Arms: Control

SUMMARY:
Peanut allergies affect approximately 2.5% of children; are associated with significant mortality, morbidity, and economic costs; and often lead to persistent peanut allergies in adulthood. We now know however that early introduction of peanut products to infants prior to age 7 months and maintained in the diet regularly significantly reduces the rate of peanut allergies. Unfortunately, recent research shows that even when parents know the recommendations to feed peanut products early and often, <50% of parents report introducing peanuts by age 9 months, <45% are offering peanut products several times a week, and <20% are offering the recommended 2 teaspoons at each feeding. Many parents cite a fear of reactions or a lack of knowledge on how to safely feed peanut products at this age. While there are recommendations to offer the first feeding in clinic this has not been widely implemented in general pediatrics clinics and we have no research to say this is an effective way to increase peanut consumption at home. This research is being conducted to assess the effectiveness of a supervised peanut feeding clinic in a pediatric office to increase rate of guideline recommended peanut consumption in infants by 9 months of age.

DETAILED DESCRIPTION:
TITLE: A Randomized Control Trial of a Supervised Peanut Feeding Clinic to Increase Early Peanut Introduction A. Specific Aims/Objectives We aim to assess if a supervised peanut feeding clinic within a general pediatrics practice can increase early peanut introduction and peanut feeding frequency by caregivers in their infants. We hypothesize that parents in the intervention arm who are offered a supervised peanut feeding clinic for their child's first feeding will be feeding peanuts more regularly at home than parents in the control arm who receive only standard guidance.

B. Background and Significance

1 in 13 children are allergic to at least one food, many are allergic to two or more, with significant associated mortality, morbidity, and economic costs1. In particular, peanut allergy is the leading pediatric food allergy in the United States, affecting ~2.5% of children2. Furthermore, approximately 83% of adults with peanut allergy report childhood onset, showing that children with peanut allergies are largely not outgrowing or being cured of this allergy3. While there are several treatments either available or in trials for curing or at least managing peanut allergy, they are expensive, time intensive, and thus not widely available4. Until recently we have had no way to prevent the onset of peanut allergy.

In 2015 the LEAP study showed that early and frequent consumption of peanut products starting by age 7 months in high-risk infants was protective against the development of a peanut allergy in childhood, with an 80% reduction in peanut allergy in those in the intervention group compared to controls who followed standard feeding guidelines at the time5. Infant feeding guidelines were changed in 2017 to recommend early peanut introduction for high-risk infants. Subsequent research has shown the benefits of early peanut introduction in all infants prompting a guideline change again in 2020 to promote early peanut introductions for all infants6,7.

Despite the robust research, the theoretical ease of implementation, and the benefits to individuals and society of guideline adherence, we continue to see low buy-in from parents. A study published in Pediatrics in 2023 by Samady and colleagues8 assessed 3062 caregivers of children ages 7 months to 3.5 years in 2021 regarding their peanut introduction habits. They stratified results by those who were aware of the guidelines; and, even amongst guideline aware parents, only 31% offered peanuts prior to 7-months with another 19.7% offering peanuts between 7-8 months. Among guideline aware parents, 8.4% offered peanuts daily or almost daily and 34.5% offered peanuts a few times a week. Finally, among guideline aware parents, reasons given for why they waited until after 7 months or did not feed at all were fear of an allergic reaction, being unaware of how to feed peanuts to an infant, and a disbelief in the guidelines.

This research shows us that while there is work to be done to ensure pediatricians are providing the guidelines to parents, guideline knowledge alone will not get us to the levels of peanut consumption in infancy that we need to make a true difference in peanut allergy prevalence. One intervention proposed in the 2017 guidelines is a supervised feeding clinic in the general pediatrician's office9 - this would address parents' fear of an allergic reaction as well as help alleviate their concerns about how to feed peanuts to an infant. However, to our knowledge no study has systematically looked at the effectiveness of offering a supervised feeding clinic. This study will look at the effect of a dedicated supervised feeding clinic on the outcome of increasing peanut introduction and consumption frequency through a randomized control trial.

C. Preliminary Studies To the best of our knowledge, there is no prior research to date specifically looking at the impact of a structured supervised peanut feeding clinic within a general pediatrics clinic setting on the rate of early peanut introduction and peanut feeding frequency in infancy.

D. Design and Methods

1. Study Design This will be an unblinded randomized control trial with two groups (Figure 1). It is not possible to blind either participants or the research team as only one group will be offered the supervised feeding clinic visit. Study team members will contact families by phone in the week after their 4-month well child visit to discuss the study and screen for eligibility. Initial information will briefly detail the goals of the study (to assess ways to help caregivers provide peanuts to their infants) and will alert them to the possibility of being assigned to the group with an extra visit, which will be billed to their insurance as a regular pediatric follow up. Caregivers who remain interested in the study will then be provided an e-consent form to enroll. All participants will receive a standard guideline handout on peanut introduction to eliminate any bias from what different pediatricians might have time to discuss with their patients and isolate the effect of the supervised feeding clinic in guideline aware caregivers. This handout is a standard guideline packet created by the Asthma and Allergy Foundation of America that is available for public use and used in our primary care clinic. Participants will then be randomized. Randomization will occur using a pre-generated block randomization chart - the chart will be twice as long as expected enrollment. The randomization determines who is offered this new resource of a supervised feeding visit, no participant is required to attend this additional visit.

   As we anticipate some caregivers will decline to participate in the study, and their reasons for doing so may inform the feasibility of offering such a clinic in the future, we will offer exit interviews for people who decline to enroll - we anticipate there might be concerns regarding transportation or visit copays related to this additional visit that we will want to assess. Families who do not wish to enroll in the RCT will be offered an opportunity to enroll in a brief qualitative interview study, anticipated to take 5 minutes, to discuss any reasons they may have had for not wanting to join the study.
2. Patient Selection and Inclusion/Exclusion Criteria All children after their 4-month well child check at our three clinical practices located at Children's Hospital Primary Care Center, Martha Eliot Health Center, and Weymouth will be assessed for eligibility. Exclusion criteria include: 1) infants who are not developmentally able to eat solids prior to age 7 months, 2) families who do not speak English, or 3) infants who have already eaten peanuts, have a positive peanut IgE (note they do not need to have a negative peanut IgE - a blood test to look for evidence of an allergy - in order to be enrolled in the study but some providers may have gotten one in their usual practice and inadvertently found a positive result), or there are other concerns regarding an existing allergy to peanuts. For any peanut allergy concerns families should be evaluated by their pediatrician and referred to Allergy & Immunology.

   Participants in the intervention arm must be at baseline state of health on the day of the supervised feeding visit, but they may be re-scheduled to another date. Unlike an oral food challenge in an Allergist's office for a known or suspected food allergy, participants in this intervention arm may have used antihistamines in the days prior to the visit. This is because this is not considered an oral food challenge, and we do not give families any such restrictions before feeding peanuts for the first time at home.
3. Description of Study Treatments or Exposures/Predictors The intervention arm will be invited to a supervised feeding clinic visit. At this clinic visit, which will take place prior to age 7 months, infants will be fed peanut butter (provided by the study team) mixed into a vehicle of choice brought by the caregivers (e.g. yogurt, cereal, mashed fruit, etc). For infants whose parents forget to bring in a mixing vehicle, we will provide apple sauce or water for thinning out the peanut butter. Feeding peanut butter itself is a minimal risk study exposure as we ask all families to do this at home by themselves without any medications or clinical team available. For this study, we are offering half the group to do what we normally ask them to do at home in the presence of a clinical team. No one in the intervention arm is required to come for this additional supervised peanut feeding visit.
4. Definition of Primary and Secondary Outcomes/Endpoints Our primary outcome is the percentage of families who have introduced peanuts by age 9 months within the home diet. Secondary outcomes include a weekly average of how often they are feeding peanut products and an average quantity fed per feeding. We will also include a balancing measure to assess if attendance at later well child visits (e.g. 9-month well child visit) is impacted by coming in for an additional visit earlier on.
5. Data Collection Methods, Assessments, Interventions and Schedule (what assessments performed, how often) All participants will receive a baseline survey after study enrollment. All participants will receive a second survey at age 9 months. Surveys were adapted from the survey used in Samady et al.8 Those in the intervention arm will be offered an in person visit to feed peanut butter to their infant in a monitored clinical setting. This visit will take place prior to age 7 months.
6. Study Timeline (as applicable) We anticipate beginning study enrollment in May 2025 and continuing through October 2025 with later enrolled participants finishing study activities in January 2026. We plan to analyze our data from January to February 2026.

E. Adverse Event Criteria and Reporting Procedures This is a minimal risk study and the study exposure - feeding peanut products to infants - is the same exposure we ask parents to do at home on their own already without medical supervision or allergic reaction treatments available. There is no new drug or supplement being investigated in this study. The only anticipated adverse event is an allergic reaction, which we expect to happen as rarely as it may occur at home (approximately <1% of the time and usually a small rash). All allergic reactions during supervised feeding visits will be documented within the clinical visit and appropriate treatment for the allergic reaction will be administered.

F. Data Management Methods All data will be stored in REDCap. G. Quality Control Method

To ensure the reliability, consistency, and safety of the study, the following quality control procedures will be implemented throughout the duration of the randomized controlled trial:

1. Randomization Process The randomization process will involve a pre-made block randomization chart which will be used for the study duration. Randomization will occur prior to any study activities.
2. Intervention Consistency

   • Clinic Visits: The intervention group will be offered a structured clinic visit, during which the baby will be examined, fed peanut butter, and then monitored for an allergic reaction. Each clinic visit will be standardized to ensure consistency in the process.
   * Standardized Feeding Protocol: ZA will administer the peanut butter with the family according to a standardized protocol. The protocol will include specific instructions on the amount of peanut butter to be given, how to safely introduce it to the baby, and any necessary monitoring for adverse reactions.
   * Supervision: The intervention will be completed by ZAwho is a pediatrician who will monitor the baby for signs of allergic reaction during the feeding and for 30 minutes afterward. Any signs of distress will be immediately addressed in accordance with the clinic's emergency procedures.
   * Documentation: Each clinic visit will be documented, including the amount of peanut butter given, any adverse reactions, and participant feedback. These records will be reviewed
3. Staff Training Only the co-investigator, Zara Rafi Atal, will be running the clinic intervention visits. She has received training through her general pediatrics practice in the correct administration of peanut butter to ensure safe feeding practices, recognition and management of allergic reactions (e.g., anaphylaxis, hives), and standardized procedures for documentation.
4. Data collection and Monitoring

   * Data Collection Tools: Standardized forms will be used for recording baseline data, clinic visit details, and follow-up data.
   * Adverse Events Monitoring: Any adverse events related to the peanut butter feeding (e.g. allergic reactions) will be documented.
5. Protocol Deviations and Corrective Actions In the event of a protocol deviation (e.g., incorrect administration of peanut butter or missed clinical visits), these will be documented, and corrective actions will be implemented. A detailed log will track all deviations and the steps taken to rectify them. The study steam will review these deviations regularly to identify trends and improve future practices.
6. Participant Feedback and Safety Checks Participants will be provided with clear instructions on what to do in case of an allergic reaction (e.g., contacting the clinic or visiting the emergency room), ensuring they have appropriate support if needed.

H. Data Analysis Plan For our primary aim we will treat our outcome as a dichotomous variable (0 = no introduction to peanuts by 9 months; 1=introduction to peanuts by 9 months). For our secondary aim we will treat our outcome as a dichotomous variable (0 = feeding peanuts 2 or fewer times a week and 1 = feeding peanuts 3 or more times per week). Our primary analysis will be an intention to treat analysis based on initial randomization group. We will run two-sample test of proportions to look at the proportion of caregivers who report at the 9-month visit that they have introduced peanuts to their infants in the intervention versus control group as well as the proportion of caregivers who report at the 9-month visit that they are giving their infant peanuts 3 or more times per week in the intervention versus control group.

Multivariable logistic regression will be used for the per-protocol analysis (comparing those who attend the supervised feeding visit to the control group) to adjust for variables that will be unbalanced once the analysis is limited to the per-protocol group.

I. Statistical Power and Sample Considerations Power calculations were done using SAS. With a sample of 58 subjects per group, we will have 80% power to detect a 50% difference in the group proportions (0.5 to 0.75) of peanut introduction prior to 9-months using a two-sided two-sample test of proportions with a significance level of 0.05. With a sample size of 80 subjects per group (of those who do introduce peanuts) we will have 80% power to detect a 50% difference in the group proportions (0.4 to 0.6) of frequency of peanut provided prior to 9-months using a two-sided two-sample test of proportions with a significance level of 0.05. To be able to test our second aim of peanut frequency and assuming a conservative 50% peanut introduction rate by the 9-month visit we will aim to enroll 160 per group. To account for a 25% loss to follow up we will aim to enroll in total 200 participants per group. Across the 3 clinics we see approximately 30 4-month well child checks per week or about 120 per month.

ELIGIBILITY:
Inclusion Criteria: All 4-6 month infants who feed by mouth who have not introduced peanuts yet and have no evidence of peanut allergy.

-

Exclusion Criteria: Non-English speaking, not eating solid food, evidence of peanut allergy.

-

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Peanut introduction at 9 months | 3 months
  Percentage of families who have introduced peanut products at home in 2 groups.

SECONDARY OUTCOMES:
Frequency of peanut introduction | 3 months
  The frequency with which families feed infants peanut products at home in two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States